CLINICAL TRIAL: NCT01607931
Title: The Effects of Acute Exercise on Glucose Kinetics, Beta-cell Function and the Incretin Effect in Subjects Representative of the Whole Glucose Tolerance Continuum
Brief Title: Exercise, Glucose Kinetics, and the Incretin Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Senior Researcher, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EFSD-2012; NCT01540097 (obsolete NCT alias)
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: Exercise; Physical activity; Type 2 diabetes; Obesity; Incretin effect; GLP-1; GIP; Insulin secretion; Glucagon; Beta-cell function; Disposition Index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resting Trial (No Intervention): a 1 hour period of rest immediately prior to OGTT or isoglycemic clamp
- Exercise Trial (Experimental): a 1 hour cycling exercise bout immediately prior to the OGTT or isoglycemic clamp
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 1 hour of cycling at 50% of maximum power output
  Arms: Exercise Trial

SUMMARY:
Human volunteers will be stratified by oral glucose tolerance status: normal glucose tolerant, impaired glucose tolerant, and type 2 diabetic. All subjects will undergo 4 experimental trials: [1] an oral glucose tolerance test (OGTT) combined with infused and ingested stable isotopes of glucose to assess glucose kinetics. [2] a 1 hour bout of cycling exercise at 50% of maximum power output, immediately followed by the same OGTT combined with stable isotope glucose tracers used in trial 1. [3] an isoglycemic clamp to match the plasma glucose profile measured in trial 1. [4] a 1 hour bout of cycling exercise at 50% of maximum power output, immediately followed by an isoglycemic clamp to match the plasma glucose profile measured in trial 2.

Exercise-induced changes in oral glucose tolerance, glucose kinetics, insulin and glucagon secretion, and the incretin effect will be examined. The exercise responses will be compared between the subjects groups of different glucose tolerance status.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* BMI 18-35 kg/m2

Exclusion Criteria:

* insulin dependency
* pregnancy
* presence or history of chronic cardiovascular, pulmonary, hepatic, renal, or hematological disease, or cancer
* contraindication to physical activity as assessed by ECG

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | Plasma glucose will be measured at 10 minute intervals during the OGTT (3 hours) immediately following the period of rest or exercise
Incretin effect | Plasma insulin and C-peptide will be measured at 10 minute intervals during the OGTT (3 hours) and isoglycemic clamp (3 hours) immediately following the period of rest or exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark